CLINICAL TRIAL: NCT05861245
Title: Phase II Clinical Trial of Low-intervention Using Hypofractionated Protontherapy in Chordomas and Chondrosarcomas of the Skull Base
Brief Title: Hypofractionated Protontherapy in Chordomas and Chondrosarcomas of the Skull Base
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Quironsalud (Other)
Responsible Party: Principal Investigator, Morena Sallabanda, MD, PhD, Quironsalud
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PIC128-22_QUIRON
Record Dates: First submitted 2023-04-26; First posted 2023-05-16 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Chordoma; Chondrosarcoma
Keywords: Skull base; Protontherapy; Hypofractionation; Chordoma; Chondrosarcoma
MeSH Terms: conditions — Chordoma; Chondrosarcoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 5 fractions (Experimental): * Patients > 18 years old.
  * With a baseline classification on the Karnofsky performance status scale ≥ 70%.
  * With confirmed histological diagnosis of chordoma or chondrosarcoma of the skull base.
  * With a maximum tumor size of 50 cc.
  * With a magnetic resonance imaging (MRI) t ruling out pre-existing vascular pathology (stenosis or atherosclerosis).
  * Whose relationship to organs at risk (OARs) allows compliance with the necessary dose restrictions to receive hypofractionated proton therapy in 5 fractions.
  Patients included in the study must meet dosimetric parameters that include:
  * Clinical Target Volume (CTV) coverage of at least D95>90%.
  * Correct compliance with the dose restrictions, at least in the nominal scenario, for critical organs (optic pathway, brain stem, spinal cord and temporal lobes) according to the guidelines published and available in the literature.
  Interventions: Radiation: 5-fraction hipofractionated protontheray
- 25 fractions (Experimental): * Patients > 18 years old.
  * With a baseline classification on the Karnofsky performance status scale ≥ 70%.
  * With confirmed histological diagnosis of chordoma or chondrosarcoma of the skull base.
  * Not considered candidates for the 5-fraction protocol due to tumor size exceeding 5 cc and/or the presence of vascular pathology identified on MRI with vascular sequences.
  * Tumor relationship to organs at risk allows compliance with the dose constraints required to receive hypofractionated proton therapy delivered in 27 fractions.
  Interventions: Radiation: 25-fraction hypofractionated proton therapy

INTERVENTIONS:
Radiation: 5-fraction hipofractionated protontheray — The therapeutic schemes that will be proposed to patients based on clinical criteria such as tumor size and relationship of the tumor with adjacent critical organs are:
  * For chordomas: 37.5 Gy in 5 consecutive sessions of 7.5 Gy per fraction.
  * For chondrosarcomas: 35 Gy in 5 consecutive sessions of 7 Gy per fraction.
  Arms: 5 fractions
Radiation: 25-fraction hypofractionated proton therapy — The therapeutic regimens to be proposed to patients, based on clinical criteria such as tumor size and the relationship between the tumor and adjacent critical organs, are as follows:
  For chordomas:
  67.5 Gy delivered in 27 consecutive fractions of 2.5 Gy per fraction to the high-risk volume, and 54 Gy delivered in 27 fractions of 2 Gy per fraction to the low-risk volume (integrated boost).
  For chondrosarcomas:
  64.8 Gy delivered in 27 consecutive fractions of 2.4 Gy per fraction to the high-risk volume, and 54 Gy delivered in 27 fractions of 2 Gy per fraction to the low-risk volume (integrated boost).
  Arms: 25 fractions

SUMMARY:
The project is planned as a phase II clinical trial with a low level of intervention, for the prospective evaluation of the clinical results of radical or adjuvant treatment by proton therapy in chordomas and chondrosarcomas of the skull base using hypofractionation schemes in 5 fractions, with the aim of consolidating the scientific evidence that exists with high-precision techniques with photons, increasing this evidence by adapting this treatment scheme to the proton technique.

In addition, a cross-sectional prospective evaluation of the quality parameters of the dosimetry of hypofractionated proton therapy and an evaluation of the quality of life of these patients will be carried out.

* Primary Objective

  1. - Toxicity according to CTCAE-v5 criteria
  2. - Local control determined by Magnetic Resonance with Gadolinium.
* Secondary Objectives

  1. To evaluate the quality of life of the patients, 3 months after the end of the treatment, using a specific questionnaire.
  2. To evaluate the dosimetric benefits using techniques that allow an improvement in the dose gradient, improving the coverage of the CTV (Clinical Tumor Volume) and decreasing the dose in surrounding risk organs.

DETAILED DESCRIPTION:
Chordomas are rare, slow-growing tumors that develop from remnants of the embryonic notochord in the clivus, sacrococcygeal region, and mobile spine. Although the frequency of distant metastases is low, these tumors are locally aggressive and have an extremely high local recurrence rate. Similarly, chondrosarcomas have a potential for slow growth with a tendency to recur locally. They usually arise at the base of the skull or spine from mesenchymal cells or from the primitive cartilaginous matrix.

Although chordomas are considered clinically more aggressive than chondrosarcomas, their tendency to settle in similar anatomical locations and the high risk of local recurrence of both diagnostic entities have conditioned a similar therapeutic approach.

Standard treatment includes surgical resection that is as radical as possible; however, complete resection is feasible in less than 50% of cases, as it can be associated with significant postoperative morbidity and mortality, since these tumors frequently invade or contact critical structures (vascular, cranial nerves or spinal roots). Therefore, adjuvant or exclusive irradiation have a fundamental role in long-term local control. Therefore, optimization of the efficacy of radiotherapy represents a critical step in the management of these patients. Given their tendency to local recurrence, chordomas require the prescription of high doses for their local control, which are associated with potentially critical adverse effects if conventional photon irradiation techniques are used.

The α/β ratio, according to the linear-quadratic model, represents a measure of the sensitivity of a tumor to variable dose-per-fraction regimens. Tumors with a low coefficient (<4 Gy) are considered more sensitive to the effects of hypofractionated treatments, which involve the administration of higher irradiation doses per session in fewer sessions.

After analyzing historical studies and institutional experiences, different publications suggest that the α/β ratio of chordomas is 2.45 Gy and it is assumed to be very similar for chondrosarcomas. Therefore, the administration of hypofractionated schedules could be associated with an increase in the sensitivity of these tumors to radiotherapy treatment.

Conventional normofractionated radiation therapy administered adjuvantly after resection has historically been used with median doses of 60 to 66.6 Gy to 2 Gy per fraction, offering 5-year local control rates ranging from 23% to 50%. Technological advances in the field of image-guided intensity-modulated radiotherapy have led to an improvement in the precision of treatments, allowing the dose for chordomas to be scaled up to 76 Gy (the biological equivalent dose (BED) taking into account the α/ β of 2.45Gy is 138 Gy) and for chondrosarcomas up to 70 Gy (BED of 127 Gy), achieving and improvement in 5-year local control rates of 65% and 88%, respectively for each diagnostic entity.

Although promising, the use of high-dose photons is limited by the lower ability to protect nearby critical organs. Therefore, particle therapy (protons and carbon ions) has established its role as a standard technique, due to its potential to achieve greater conformation and better dose distribution. The main studies with proton therapy for these tumors appear to show statistically significant results in favor of increased survival when dose escalation above 70 Gy to 2 Gy per fraction (BED >127 Gy) is compared with techniques using irradiation with intensity modulated photons (IMRT). The 5-year local control rate is above 60% for chordomas and above 80% for chondrosarcomas with moderate toxicity and preservation of critical structures. However, the limited availability of these facilities together with the administration of very long treatment schedules, often of seven weeks or more, poses a significant problem for patients and remains an obstacle to the widespread adoption of this technique as a therapeutic standard.

Due to all these limitations and the important advances in terms of precision and dose distribution, the concept of hypofractionation has gained weight within radiation oncology thanks to its potential benefits in terms of reducing the duration of treatment and costs. The first publications on the hypofractionated treatment of chordomas, mainly of the skull base, go hand in hand with photon radiosurgery systems, using dedicated equipment such as the GammaKnife or CyberKnife. In the last 15 years, single-dose or hypofractionated treatment schemes have been explored as a therapeutic alternative to escalate the dose, improve the protection of organs at risk and reduce treatment time.

Some studies have evaluated single fraction stereotactic radiosurgery (SRS) in the management of chordomas and chondrosarcomas mainly located in the skull base with results comparable to proton therapy. The most relevant studies included series of 22 to 71 patients treated with median doses of SRS ranging from 12.7-24 Gy (BED 78.5-259 Gy). Five-year local control rates ranged from 21-85%, depending on the doses prescribed (higher doses, ≥15 Gy, were associated with better relapse-free survival).

However, based on the experience of Kano et al., for single-dose treatments, irradiation of volumes > 7 cc is associated with a significant worsening of tumor control. It is essential to emphasize that the tumor volumes that are usually treated in chordomas and chondrosarcomas, both at the base of the skull and, to a greater extent, in the spine, exceed, in most cases, 7 cc, since the entire clivus or affected vertebral bodies must be included in the majority of cases, in order to reduce the risk of marginal recurrence. For this reason, the role of single-dose radiosurgery loses weight in favor of hypofractionated stereotactic radiotherapy (HFSRT), which has theoretical advantages compared to single-dose treatment in volumes greater than 7 cc, including a lower risk of radiation-induced toxicity in nearby critical structures and the possibility of safely treating larger tumor volumes with multiple fractions (usually 5).

Several publications evaluate HFSRT for chordomas and chondrosarcomas. The number of cases included in these series ranged from 9 to 24 patients. The median follow-up was 24 to 46 months. Most patients were treated with 5 fractions with a prescription dose of 24-43 Gy (BED 52.7-194 Gy), depending on histology and therapeutic setting (radical, adjuvant, or reirradiation). The best local control results at 3 and 5 years obtained were 90 and 60% for chordomas, respectively, and 100% for chondrosarcomas. The most widely used regimen was 37.5 Gy in 5 fractions of 7.5 Gy (BED 152.3 Gy equivalent to 80 Gy at 2 Gy per fraction) for chordomas and 35 Gy in 5 fractions of 7 Gy per fraction in Chondrosarcomas (BED of 135 Gy equivalent to 74 Gy at 2 Gy per fraction). The toxicity described in most of these studies does not register worse data than those published with conventional fractionation in proton therapy, when it comes to primary treatments.

This growing evidence, which is described as a justification for the implementation of hypofractionated regimens, demonstrates that the standard implementation of these therapeutic modalities in patients who meet the appropriate characteristics can suppose a great advantage to improve accessibility and comfort for patients, potentially reduce acute side effects during treatment and increase therapeutic cost-efficiency.

Proton therapy, today, remains a limited resource, with only 99 facilities currently in operation worldwide in 2021, of which two new centers are in Spain, active since 2020. In addition, many patients must travel to access to this technology, so reducing the time a patient is away from home and their support network can have significant financial and psychosocial implications. Added to all this are the aforementioned radiobiological advantages of high doses per fraction, in tumors with a low α/β coefficient, such as chordomas and chondrosarcomas. That is why the implementation of hypofractionation within proton therapy has gained weight in the last 10 years, increasing the number of publications in this regard, which reflects the interest in this treatment approach.

Cao et al. presented a dosimetric study comparing different hypofractionated stereotactic treatment schemes in the treatment of intracranial tumors > 3 cm in greatest diameter. Treatment plans with GammaKnife, Cyberknife and VMAT were generated compared with proton therapy plans with or without modulated intensity. The authors suggest that proton therapy represents a desirable alternative to advanced photon techniques for treating large, irregularly shaped volumes near critical structures, such as chordomas and chondrosarcomas.

For all these reasons, a fundamental and necessary challenge today consists of increasing the scientific evidence of hypofractionated schemes in the treatment of chordomas and chondrosarcomas, adapting them to protontherapy, to increase clinical experience and combine the benefits of high-precision hypofractionated treatments to the dosimetric advantages of protontherapy (ability to treat volumes > 7 cc with a homogeneity index close to 1 and a decrease in the integral dose in healthy tissue).

In summary, considering the growing scientific evidence available from other studies on different therapeutic entities, we have a solid basis to reinforce hypofractionation protocols with protontherapy in the treatment of chordomas and chondrosarcomas.

The main advantages of these protocols, as mentioned above, are aimed at optimizing the treatment of these patients by providing potential clinical benefits derived from the advantages associated with the biological response to high doses per fraction, reducing the likelihood of acute side effects, increasing the availability and accessibility of proton therapy units to a larger number of patients, and optimizing therapeutic cost-effectiveness.

As disadvantages, these protocols are intended for a limited subgroup of patients who meet strict criteria, including small-volume lesions located at the skull base and sufficiently distant from organs at risk that are sensitive to high doses per fraction, such as the brainstem and the optic pathway, in order to avoid the development of potentially disabling chronic side effects.

Based on all of the above, we decided to design a first prospective study which, with the support and recommendations of this committee, became a clinical trial entitled: "Low-intervention Clinical Trial of Hypofractionated Proton Therapy in Skull Base Chordomas and Chondrosarcomas", approved on 26/09/2023 (PIC128_22_QUIRON). We published our initial results from the prospective series, which included 11 patients treated using the same criteria applied in the clinical trial, along with a description of the trial. Since its approval, three patients have been recruited within the clinical trial, resulting in a total of 14 patients treated under the same conditions, with a median follow-up of 28 months.

Based on the follow-up data obtained, we decided to perform an interim analysis to evaluate outcomes. Local control was 100% throughout the entire follow-up period. One patient died from complications secondary to treatments 32 months after proton therapy (reoperation for basilar artery stenosis and cerebrospinal fluid fistula following surgery). Acute tolerance was excellent in all patients; however, regarding chronic toxicity, we observed a higher number of temporal lobe necrosis cases than initially described in normofractionated proton therapy series, occurring between 8 months and 2 years after treatment administration (median of 12 months after proton therapy).

Five patients were diagnosed with radiological radionecrosis (35.7% of the series, compared with 15% reported in the literature for normofractionated regimens) (39). Of these, three presented symptoms clearly related to imaging findings: in two patients, symptoms were mild and resolved with corticosteroid therapy (grade I-II asthenia, grade I-II headache, and a single isolated seizure episode). In another patient, symptoms were more severe (seizures and memory impairment) and were associated with other post-surgical complications (basilar artery stenosis), which ultimately led to the patient's death. The factor most clearly associated with the higher incidence of radionecrosis appears to be the maximum dose received by the affected temporal lobes (greater than 34 Gy in 2% of the volume).

The greater the risk of creating "hot spots," the higher the predisposition of the local vasculature surrounding the target to increased vascular injury, one of the potential triggers of radionecrosis. Changes in microvascular permeability and loss of blood-brain barrier integrity are key features of radiation-induced injury in the central nervous system, as is the expression of vascular endothelial growth factor (VEGF). Inherent to the nature of particle beams, proton therapy exhibits greater relative biological effectiveness (RBE) than photon-based radiotherapy, which may increase the risk of radionecrosis and subsequently enhance the inflammatory response and vasculopathy. This effect is explained by a higher linear energy transfer (LET), resulting in greater local energy deposition. DNA damage increases in quantity and/or complexity, representing a greater burden on the cellular repair system. This increased efficacy of ionizing radiation is quantified as the RBE. Numerous studies have demonstrated a clear increase in RBE toward the Bragg peak, where protons stop (at the end of the beam) and where LET is comparatively high.

Histologically, radiation-induced brain necrosis is characterized by the presence of geographic eosinophilic necrosis accompanied by gemistocytic astrocytes representing gliosis with atypia. In addition, fibrinoid vascular necrosis associated with dystrophic calcification, perivascular lymphoplasmacytic infiltrates, and telangiectasias representing reactive vascular changes are also observed, although these findings are not highly specific to radiation-induced brain necrosis. There is significant interpatient variability in radiosensitivity. Initial evidence supporting a genetic basis for radiation toxicity came from studies in breast cancer patients, in whom approximately 90% of the variation in the development of radiation-induced telangiectasia was attributed to underlying genetic differences. Patients with ataxia-telangiectasia, Fanconi anemia, and Bloom syndrome-hereditary disorders involving DNA damage surveillance and repair genes-exhibit increased radiosensitivity. The diverse genetic abnormalities responsible for these disorders suggest that radiosensitivity is polygenic, involving multiple pathways, some of which are inherited. In recent years, a broader genome-wide approach has been adopted. A recent genome-wide association study revealed a variable risk of radiation-induced temporal lobe necrosis associated with different single-nucleotide polymorphisms in a glioblastoma cell line (U87) treated with X-rays and H₂O₂. This is the first study implicating a susceptibility gene for radiation injury (Cep128) and provides novel insights into the underlying mechanisms of radiation-induced brain injury.

Based on the above, we believe that the increased rates of radionecrosis have a multifactorial component. On the one hand, there may be a greater predisposition to vascular damage, potentially related to pre-existing vascular injury prior to treatment (tumoral, post-surgical, or hereditary). Furthermore, in skull base tumors such as chordomas and chondrosarcomas, the distal end of the beams is often oriented toward the temporal lobes in order to avoid more sensitive structures such as the optic pathway or the brainstem, thereby increasing LET and RBE in this location. This enhances the radiobiological effect which, together with the increased dose per fraction, could explain the higher incidence of temporal lobe necrosis.

For all these reasons, we would like to request a protocol amendment to optimize inclusion criteria and improve planning quality parameters, with the aim of reducing the risk of temporal lobe radionecrosis while allowing patients to benefit from the advantages of improved acute tolerance, reduced treatment duration, and improved local control. For patients who are not candidates for extreme hypofractionation schemes (5 fractions), we will add a moderately hypofractionated arm with an integrated boost protocol (27 fractions).

In summary, the research project is based on the performance of a phase II clinical trial with a low level of intervention, which consists of the prospective evaluation of the clinical and radiological response after the administration of a treatment using radical or adjuvant hypofractionated proton therapy in 5 or 27 sessions in patients diagnosed with chordoma or chondrosarcoma of the skull base.

In addition, a cross-sectional evaluation of the quality parameters of the dosimetry of the hypofractionated proton therapy treatments administered to the patients included in the study and an evaluation of the quality of life by means of specific questionnaires, 3 months after treatment, will be carried out.

ELIGIBILITY:
Inclusion Criteria for 5 fractions:

* With a baseline classification on the Karnofsky performance status scale ≥ 70%.
* With confirmed histological diagnosis of chordoma or chondrosarcoma of the skull base.
* Who have signed the specific informed consent of the protocol, agreeing to participate in it.
* Completion of magnetic resonance imaging with vascular assessment ruling out pre-existing vascular pathology (stenosis or atherosclerosis), including 3D T1 black-blood sequences, pre-contrast 3D TOF, 3D T2 with fat suppression, and perfusion sequences.
* With a maximum tumor size of 50 cc.
* Whose relationship to organs at risk (OARs) allows compliance with the necessary dose restrictions to receive hypofractionated proton therapy in 5 fractions.
* Patients included in the study must meet dosimetric parameters that include:
* Tumor CTV coverage of at least D95>90%.
* Correct compliance with the dose restrictions, at least in the nominal scenario, for critical organs (optic pathway, brain stem and spinal cord) according to the guidelines published and available in the literature:

Dose contnstraints for 5 fractions:

Optic Nerves: D0.03cc ≤ 25 GyRBE, V23.5 < 0.5cc. Chiasm:D0.03cc ≤ 25 GyRBE, V23.5 < 0.5cc. Brainstem:D0.03cc ≤ 31 GyRBE,V23 < 0.5cc. Spinal Chord: D0.03cc ≤ 30 GyRBE, V23 < 035cc. Right and left temporal lobes: D0.03 cc ≤ 35 GyRBE, V30 ≤ 5.5 cc.

Inclusion Criteria for 25 fractions:

* With a baseline classification on the Karnofsky performance status scale ≥ 70%.
* With confirmed histological diagnosis of chordoma or chondrosarcoma of the skull base.
* Who have signed the specific informed consent of the protocol, agreeing to participate in it.
* Not considered candidates for the 5-fraction protocol due to tumor size exceeding 50 cc and/or the presence of vascular pathology (stenosis or atherosclerosis) identified on MRI with vascular sequences.
* Tumor relationship to organs at risk allows compliance with the dose constraints required to receive hypofractionated proton therapy delivered in 27 fractions.
* Patients included in the study must meet dosimetric parameters that include:
* Tumor CTV coverage of at least D95>90%.
* Correct compliance with the dose restrictions, at least in the nominal scenario, for critical organs (optic pathway, brain stem and spinal cord) according to the guidelines published and available in the literature:

Dose constraints for 25 fractions:

Optic nerves: D0.03 cc ≤ 54.7 GyRBE. Optic chiasm: D0.03 cc ≤ 54.7 GyRBE. Brainstem: Surface: D0.03 cc ≤ 57.9 GyRBE. Core: D0.03 cc ≤ 54 GyRBE. Spinal cord: D0.03 cc ≤ 54 GyRBE. Right and left temporal lobes: V65 < 1.7 cc, V60 ≤ 5.5 cc.

Treatment planning with a minimum of 5 beams. In general, the use of a class solution with 6 beams will be proposed, including 2 lateral beams with gantry angles between 20° and 80°, depending on tumor location; 2 posterior oblique beams; and 2 anterior oblique beams. The latter four beams may include a couch rotation of at least 20° relative to the two lateral beams, with a minimum angular separation of at least 30° between ipsilateral oblique beams. Depending on individual patient characteristics, this class solution will be adapted to adjust specific gantry and couch angles for each field.

If this solution is not feasible due to patient-specific characteristics (surgical constraints, tumor location or laterality, etc.), a 5-beam solution will be evaluated, including 2 posterior oblique beams and 2 anterior oblique beams, in addition to a coronal field with the couch at 270° and a gantry angle between 40° and 90° depending on tumor location, or other configurations that increase the number of ipsilateral oblique beams with a minimum inter-beam separation of at least 30°.

Evaluation of Linear Energy Transfer (LET) and biological dose:

For each treatment plan, the LET distribution obtained from the treatment planning system (TPS) will be evaluated, with particular attention to regions where LET values exceed 5 keV/μm, aiming to minimize such values. Equivalent biological dose distributions based on recognized models in the literature may also be assessed to support decision-making regarding the suitability of a given treatment plan

Exclusion Criteria:

* Patients with distant metastases.
* Patients who have received previous irradiation in the same location.
* Patients whose clinical or dosimetric characteristics do not meet the inclusion criteria.
* Patients who are simultaneously participating in another study that may affect the results of this protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2023-05-24 (Actual); Primary Completion 2027-05-24 (Estimated); Study Completion 2033-05-24 (Estimated)

PRIMARY OUTCOMES:
Acute treatment tolerance | 0 - 3 months
  To evaluate acute toxicity using the Common Terminology Criteria for Adverse Events (CTCAE) scale, of the implementation of hypofractionation schemes in the treatment with protontherapy of skull base chordomas and chondrosarcomas.
Chronic treatment tolerance | 3 months - 10 years
  To evaluate chronic toxicity using the Common Terminology Criteria for Adverse Events (CTCAE) scale, of the implementation of hypofractionation schemes in the treatment with protontherapy of skull base chordomas and chondrosarcomas.
Local control | 1 - 10 years
  To evaluate the clinical impact in terms of local control based on the radiological findings by MRI with gadolinium (considering progression to an increase in tumor volume > 10%).

SECONDARY OUTCOMES:
Quality of life after treatment - QLQ-C30 | 3 months
  To evaluate the quality of life of the patients included in the study, for this, in a period of 3 months after the end of treatment, the patients will be summoned in person at the center to carry out the questionnaire of quality of life for cancer patients EORTC QLQ-C30.
Quality of life after treatmenT- QLQ-BN20 | 3 months
  To evaluate the quality of life of the patients included in the study, for this, in a period of 3 months after the end of treatment, the patients will be summoned in person at the center to carry out the questionnaire of quality of life for cancer patients with central nervous system tumors, EORTC QLQ-BN20.
Dosimetric benefits | 3 months
  To evaluate the dosimetric benefits using techniques that allow an improvement in the dose gradient, improving the coverage of the CTV (Clinical Tumor Volume) and decreasing the dose in surrounding risk organs. For this, apertures will be used whenever necessary to reduce the dose in surrounding tissues and the pre-treatment dosimetric distributions will be verified.

CONTACTS AND LOCATIONS:
Locations (1):
- Centro de Protonterapia Quironsalud, Madrid, Madrid, Spain

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Ali FS, Arevalo O, Zorofchian S, Patrizz A, Riascos R, Tandon N, Blanco A, Ballester LY, Esquenazi Y. Cerebral Radiation Necrosis: Incidence, Pathogenesis, Diagnostic Challenges, and Future Opportunities. Curr Oncol Rep. 2019 Jun 19;21(8):66. doi: 10.1007/s11912-019-0818-y. PMID 31218455
- [Background] Friedrich T. Proton RBE dependence on dose in the setting of hypofractionation. Br J Radiol. 2020 Mar;93(1107):20190291. doi: 10.1259/bjr.20190291. Epub 2019 Aug 28. PMID 31437004
- [Background] McDonald MW, Linton OR, Moore MG, Ting JY, Cohen-Gadol AA, Shah MV. Influence of Residual Tumor Volume and Radiation Dose Coverage in Outcomes for Clival Chordoma. Int J Radiat Oncol Biol Phys. 2016 May 1;95(1):304-311. doi: 10.1016/j.ijrobp.2015.08.011. Epub 2015 Aug 7. PMID 26519991
- [Background] Sallabanda M, Vera JA, Perez JM, Matute R, Montero M, de Pablo A, Cerron F, Valero M, Castro J, Mazal A, Miralbell R. Five-Fraction Proton Therapy for the Treatment of Skull Base Chordomas and Chondrosarcomas: Early Results of a Prospective Series and Description of a Clinical Trial. Cancers (Basel). 2023 Nov 25;15(23):5579. doi: 10.3390/cancers15235579. PMID 38067283
- [Background] Bakker SH, Jacobs WCH, Pondaag W, Gelderblom H, Nout RA, Dijkstra PDS, Peul WC, Vleggeert-Lankamp CLA. Chordoma: a systematic review of the epidemiology and clinical prognostic factors predicting progression-free and overall survival. Eur Spine J. 2018 Dec;27(12):3043-3058. doi: 10.1007/s00586-018-5764-0. Epub 2018 Sep 15. PMID 30220042
- [Background] Walcott BP, Nahed BV, Mohyeldin A, Coumans JV, Kahle KT, Ferreira MJ. Chordoma: current concepts, management, and future directions. Lancet Oncol. 2012 Feb;13(2):e69-76. doi: 10.1016/S1470-2045(11)70337-0. PMID 22300861
- [Background] Gelderblom H, Hogendoorn PC, Dijkstra SD, van Rijswijk CS, Krol AD, Taminiau AH, Bovee JV. The clinical approach towards chondrosarcoma. Oncologist. 2008 Mar;13(3):320-9. doi: 10.1634/theoncologist.2007-0237. PMID 18378543
- [Background] Jiang B, Veeravagu A, Feroze AH, Lee M, Harsh GR, Soltys SG, Gibbs IC, Adler JR, Chang SD. CyberKnife radiosurgery for the management of skull base and spinal chondrosarcomas. J Neurooncol. 2013 Sep;114(2):209-18. doi: 10.1007/s11060-013-1172-9. Epub 2013 Jun 8. PMID 23748573
- [Background] Austin JP, Urie MM, Cardenosa G, Munzenrider JE. Probable causes of recurrence in patients with chordoma and chondrosarcoma of the base of skull and cervical spine. Int J Radiat Oncol Biol Phys. 1993 Feb 15;25(3):439-44. doi: 10.1016/0360-3016(93)90065-4. PMID 8436522
- [Background] Bohman LE, Koch M, Bailey RL, Alonso-Basanta M, Lee JY. Skull base chordoma and chondrosarcoma: influence of clinical and demographic factors on prognosis: a SEER analysis. World Neurosurg. 2014 Nov;82(5):806-14. doi: 10.1016/j.wneu.2014.07.005. Epub 2014 Jul 5. PMID 25009165
- [Background] Vasudevan HN, Raleigh DR, Johnson J, Garsa AA, Theodosopoulos PV, Aghi MK, Ames C, McDermott MW, Barani IJ, Braunstein SE. Management of Chordoma and Chondrosarcoma with Fractionated Stereotactic Radiotherapy. Front Surg. 2017 Jun 23;4:35. doi: 10.3389/fsurg.2017.00035. eCollection 2017. PMID 28691010
- [Background] Crockard A. Chordomas and chondrosarcomas of the cranial base: results and follow-up of 60 patients. Neurosurgery. 1996 Feb;38(2):420. doi: 10.1097/00006123-199602000-00044. No abstract available. PMID 8869078
- [Background] Gwak HS, Yoo HJ, Youn SM, Chang U, Lee DH, Yoo SY, Rhee CH. Hypofractionated stereotactic radiation therapy for skull base and upper cervical chordoma and chondrosarcoma: preliminary results. Stereotact Funct Neurosurg. 2005;83(5-6):233-43. doi: 10.1159/000091992. Epub 2006 Mar 13. PMID 16601376
- [Background] Amendola BE, Amendola MA, Oliver E, McClatchey KD. Chordoma: role of radiation therapy. Radiology. 1986 Mar;158(3):839-43. doi: 10.1148/radiology.158.3.3945761.
- [Background] Tai PT, Craighead P, Bagdon F. Optimization of radiotherapy for patients with cranial chordoma. A review of dose-response ratios for photon techniques. Cancer. 1995 Feb 1;75(3):749-56. doi: 10.1002/1097-0142(19950201)75:33.0.co;2-d. PMID 7828124
- [Background] Thames HD, Suit HD. Tumor radioresponsiveness versus fractionation sensitivity. Int J Radiat Oncol Biol Phys. 1986 Apr;12(4):687-91. doi: 10.1016/0360-3016(86)90081-7. PMID 3700173
- [Background] Henderson FC, McCool K, Seigle J, Jean W, Harter W, Gagnon GJ. Treatment of chordomas with CyberKnife: georgetown university experience and treatment recommendations. Neurosurgery. 2009 Feb;64(2 Suppl):A44-53. doi: 10.1227/01.NEU.0000341166.09107.47. PMID 19165073
- [Background] Sallabanda M, Garcia R, Lorenzana L, Santaolalla I, Abarca J, Sallabanda K. Treatment of Chordomas and Chondrosarcomas With CyberKnife Robotic Hypofractionated Radiosurgery: A Single Institution Experience. Cureus. 2021 Aug 8;13(8):e17012. doi: 10.7759/cureus.17012. eCollection 2021 Aug. PMID 34405079
- [Background] Kilby W, Dooley JR, Kuduvalli G, Sayeh S, Maurer CR Jr. The CyberKnife Robotic Radiosurgery System in 2010. Technol Cancer Res Treat. 2010 Oct;9(5):433-52. doi: 10.1177/153303461000900502. PMID 20815415
- [Background] Fuchs B, Dickey ID, Yaszemski MJ, Inwards CY, Sim FH. Operative management of sacral chordoma. J Bone Joint Surg Am. 2005 Oct;87(10):2211-6. doi: 10.2106/JBJS.D.02693. PMID 16203885
- [Background] Palm RF, Oliver DE, Yang GQ, Abuodeh Y, Naghavi AO, Johnstone PAS. The role of dose escalation and proton therapy in perioperative or definitive treatment of chondrosarcoma and chordoma: An analysis of the National Cancer Data Base. Cancer. 2019 Feb 15;125(4):642-651. doi: 10.1002/cncr.31958. Epub 2019 Jan 14. PMID 30644538
- [Background] Pamir MN, Kilic T, Ture U, Ozek MM. Multimodality management of 26 skull-base chordomas with 4-year mean follow-up: experience at a single institution. Acta Neurochir (Wien). 2004 Apr;146(4):343-54; discusion 354. doi: 10.1007/s00701-004-0218-3. Epub 2004 Feb 16. PMID 15057528
- [Background] Bloch OG, Jian BJ, Yang I, Han SJ, Aranda D, Ahn BJ, Parsa AT. A systematic review of intracranial chondrosarcoma and survival. J Clin Neurosci. 2009 Dec;16(12):1547-51. doi: 10.1016/j.jocn.2009.05.003. Epub 2009 Sep 30. PMID 19796952
- [Background] Zorlu F, Gurkaynak M, Yildiz F, Oge K, Atahan IL. Conventional external radiotherapy in the management of clivus chordomas with overt residual disease. Neurol Sci. 2000 Aug;21(4):203-7. doi: 10.1007/s100720070077. PMID 11214658
- [Background] Sahgal A, Chan MW, Atenafu EG, Masson-Cote L, Bahl G, Yu E, Millar BA, Chung C, Catton C, O'Sullivan B, Irish JC, Gilbert R, Zadeh G, Cusimano M, Gentili F, Laperriere NJ. Image-guided, intensity-modulated radiation therapy (IG-IMRT) for skull base chordoma and chondrosarcoma: preliminary outcomes. Neuro Oncol. 2015 Jun;17(6):889-94. doi: 10.1093/neuonc/nou347. Epub 2014 Dec 27. PMID 25543126
- [Background] Fossati P, Vavassori A, Deantonio L, Ferrara E, Krengli M, Orecchia R. Review of photon and proton radiotherapy for skull base tumours. Rep Pract Oncol Radiother. 2016 Jul-Aug;21(4):336-55. doi: 10.1016/j.rpor.2016.03.007. Epub 2016 Apr 16. PMID 27330419
- [Background] DeLaney TF, Liebsch NJ, Pedlow FX, Adams J, Dean S, Yeap BY, McManus P, Rosenberg AE, Nielsen GP, Harmon DC, Spiro IJ, Raskin KA, Suit HD, Yoon SS, Hornicek FJ. Phase II study of high-dose photon/proton radiotherapy in the management of spine sarcomas. Int J Radiat Oncol Biol Phys. 2009 Jul 1;74(3):732-9. doi: 10.1016/j.ijrobp.2008.08.058. Epub 2008 Dec 25. PMID 19095372
- [Background] Ares C, Hug EB, Lomax AJ, Bolsi A, Timmermann B, Rutz HP, Schuller JC, Pedroni E, Goitein G. Effectiveness and safety of spot scanning proton radiation therapy for chordomas and chondrosarcomas of the skull base: first long-term report. Int J Radiat Oncol Biol Phys. 2009 Nov 15;75(4):1111-8. doi: 10.1016/j.ijrobp.2008.12.055. Epub 2009 Apr 20. PMID 19386442
- [Background] Indelicato DJ, Rotondo RL, Begosh-Mayne D, Scarborough MT, Gibbs CP, Morris CG, Mendenhall WM. A Prospective Outcomes Study of Proton Therapy for Chordomas and Chondrosarcomas of the Spine. Int J Radiat Oncol Biol Phys. 2016 May 1;95(1):297-303. doi: 10.1016/j.ijrobp.2016.01.057. PMID 27084648
- [Background] Liu AL, Wang ZC, Sun SB, Wang MH, Luo B, Liu P. Gamma knife radiosurgery for residual skull base chordomas. Neurol Res. 2008 Jul;30(6):557-61. doi: 10.1179/174313208X297878. PMID 18647493
- [Background] Kano H, Iqbal FO, Sheehan J, Mathieu D, Seymour ZA, Niranjan A, Flickinger JC, Kondziolka D, Pollock BE, Rosseau G, Sneed PK, McDermott MW, Lunsford LD. Stereotactic radiosurgery for chordoma: a report from the North American Gamma Knife Consortium. Neurosurgery. 2011 Feb;68(2):379-89. doi: 10.1227/NEU.0b013e3181ffa12c. PMID 21135744
- [Background] Iyer A, Kano H, Kondziolka D, Liu X, Niranjan A, Flickinger JC, Lunsford LD. Stereotactic radiosurgery for intracranial chondrosarcoma. J Neurooncol. 2012 Jul;108(3):535-42. doi: 10.1007/s11060-012-0858-8. Epub 2012 Apr 11. PMID 22492245
- [Background] Kano H, Sheehan J, Sneed PK, McBride HL, Young B, Duma C, Mathieu D, Seymour Z, McDermott MW, Kondziolka D, Iyer A, Lunsford LD. Skull base chondrosarcoma radiosurgery: report of the North American Gamma Knife Consortium. J Neurosurg. 2015 Nov;123(5):1268-75. doi: 10.3171/2014.12.JNS132580. Epub 2015 Jun 26. PMID 26115468
- [Background] Yamada Y, Laufer I, Cox BW, Lovelock DM, Maki RG, Zatcky JM, Boland PJ, Bilsky MH. Preliminary results of high-dose single-fraction radiotherapy for the management of chordomas of the spine and sacrum. Neurosurgery. 2013 Oct;73(4):673-80; discussion 680. doi: 10.1227/NEU.0000000000000083. PMID 23842548
- [Background] Jiang B, Veeravagu A, Lee M, Harsh GR, Lieberson RE, Bhatti I, Soltys SG, Gibbs IC, Adler JR, Chang SD. Management of intracranial and extracranial chordomas with CyberKnife stereotactic radiosurgery. J Clin Neurosci. 2012 Aug;19(8):1101-6. doi: 10.1016/j.jocn.2012.01.005. Epub 2012 Jun 20. PMID 22727205
- [Background] Santos A, Penfold S, Gorayski P, Le H. The Role of Hypofractionation in Proton Therapy. Cancers (Basel). 2022 May 2;14(9):2271. doi: 10.3390/cancers14092271. PMID 35565400
- [Background] Cao H, Xiao Z, Zhang Y, Kwong T, Danish SF, Weiner J, Wang X, Yue N, Dai Z, Kuang Y, Bai Y, Nie K. Dosimetric comparisons of different hypofractionated stereotactic radiotherapy techniques in treating intracranial tumors > 3 cm in longest diameter. J Neurosurg. 2019 Mar 22;132(4):1024-1032. doi: 10.3171/2018.12.JNS181578. Print 2020 Apr 1. PMID 30901747
- [Background] Timmerman R. A Story of Hypofractionation and the Table on the Wall. Int J Radiat Oncol Biol Phys. 2022 Jan 1;112(1):4-21. doi: 10.1016/j.ijrobp.2021.09.027. No abstract available. PMID 34919882
- [Background] Diez P, Hanna GG, Aitken KL, van As N, Carver A, Colaco RJ, Conibear J, Dunne EM, Eaton DJ, Franks KN, Good JS, Harrow S, Hatfield P, Hawkins MA, Jain S, McDonald F, Patel R, Rackley T, Sanghera P, Tree A, Murray L. UK 2022 Consensus on Normal Tissue Dose-Volume Constraints for Oligometastatic, Primary Lung and Hepatocellular Carcinoma Stereotactic Ablative Radiotherapy. Clin Oncol (R Coll Radiol). 2022 May;34(5):288-300. doi: 10.1016/j.clon.2022.02.010. Epub 2022 Mar 7. PMID 35272913
- [Background] Grimm J, LaCouture T, Croce R, Yeo I, Zhu Y, Xue J. Dose tolerance limits and dose volume histogram evaluation for stereotactic body radiotherapy. J Appl Clin Med Phys. 2011 Feb 8;12(2):3368. doi: 10.1120/jacmp.v12i2.3368. PMID 21587185
- [Background] Freites-Martinez A, Santana N, Arias-Santiago S, Viera A. Using the Common Terminology Criteria for Adverse Events (CTCAE - Version 5.0) to Evaluate the Severity of Adverse Events of Anticancer Therapies. Actas Dermosifiliogr (Engl Ed). 2021 Jan;112(1):90-92. doi: 10.1016/j.ad.2019.05.009. Epub 2020 Sep 3. No abstract available. English, Spanish. PMID 32891586